CLINICAL TRIAL: NCT04958343
Title: Application and Clinical Effectiveness of Pelvic Reconstruction in Robot-assisted Radical Cystectomy-orthotopic Ileal Neobladder in the Male
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SysMU-RARC4
Record Dates: First submitted 2021-07-09; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- reconstruction group: Patients will receive pelvic reconstruction following radical cystectomy during the operation.
  Interventions: Procedure: pelvic reconstruction
- non-reconstruction group: Patients will not receive pelvic reconstruction following radical cystectomy during the operation.

INTERVENTIONS:
Procedure: pelvic reconstruction — After radical cystectomy, the pelvic reconstruction including the ligation of dorsal vascular complex and posterior reconstruction will be performed on patients.
  Groups: reconstruction group

SUMMARY:
To study the effect of pelvic reconstruction on early return of continence after robot-assisted radical cystectomy-orthotopic ileal neobladder in the male.

DETAILED DESCRIPTION:
This study will enroll male patients with bladder cancer who will undergo robot-assisted radical cystectomy-orthotopic ileal neobladder. The patients will be distributed into two comparable groups according to whether received pelvic reconstruction or not. Patient demographics and pathologic, perioperative, functional, and oncologic outcomes will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 18 or older.
2. Patients those who are diagnosed with urothelial carcinoma.
3. Patients those who are capable of receiving radical cystectomy with orthotopic ileal neobladder.
4. Patients those who are able to cooperate and complete the follow-up.
5. Patients those who volunteer to participate in this study and sign the informed consens.

Exclusion Criteria:

1. Patients thsoe who are diagnosed distant metastasis before surgery.
2. Patients those who are diagnosed with other malignancies.
3. Patients those who had received pelvic radiotherapy or major pelvic operation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enroll patients who received RARC.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-02 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
day-time and night-time continence rate | 6 months
  Patients were considered continent when they required 0 or 1 safety pad during the day or at night.

SECONDARY OUTCOMES:
perioperative complication rate | 3 months
operative time | 24 hours
estimated blood loss | 24 hours
overall survival | 1 year
recurrence-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No